CLINICAL TRIAL: NCT06742775
Title: Evolution of the Relationship Between Central and Peripheral Arterial Wave Velocities as a Function of Age
Acronym: EvolVOAge
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Grenoble Alps (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0299
Record Dates: First submitted 2024-12-11; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Aging; Diagnostic Techniques, Cardiovascular
Keywords: photoplethysmography; electrocardiography; inductive plethysmography; Pulse Wave Velocity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Under 30: Healthy volunteers younger than 30 years
  Interventions: Other: physiological signal acquisitions
- Between 30 and 50: Healthy volunteers between 30 and 50 years
  Interventions: Other: physiological signal acquisitions
- More than 50: Healthy volunteers older than 50 years
  Interventions: Other: physiological signal acquisitions

INTERVENTIONS:
Other: physiological signal acquisitions — Subjects will be fitted with non-intrusive devices. In a semi-recumbent position, they will be asked to perform
  * 10 minutes of resting breathing
  * 10 cycles consisting of a 20-second apnea, to be performed at the end of inspiration, and 1 minute 40 of breathing (100 seconds).
  This single participation session will last a total of one hour for the volunteer (equipment, recording, de-equipping), including 30 minutes of acquisition.

SUMMARY:
Acquisition of synchronized cardiovascular signals from non-invasive measurements (ECG, photoplethysmography pulse sensors, inductance plethysmography) in healthy volunteers aged from 18 to 75, during spontaneous ventilation with apneas (20 seconds) for a total acquisition time of 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 75 years of age
* No acute cardiovascular pathologies less than 2 years old,
* No chronic cardiovascular pathologies.
* Stature compatible with the use of the plethysmography T-shirt.
* Person affiliated to a social security scheme or beneficiary of such a scheme
* Signed informed consent form

Exclusion Criteria:

* Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care under articles L. 3212-1 and L. 3213-1 who are not covered by the provisions of article L. 1121-8, persons admitted to a health or social establishment for purposes other than research, minors, persons under legal protection or unable to express their consent).
* Personnel with a hierarchical link to the principal investigator
* Subjects excluded from another study,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 60 healthy volunteers: 3 groups of 20 volunteers per age category (under 30, between 30 and 50, over 50)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Electrocardiogram | 1 hour
  acquisition of ECG signals
Photoplethysmography | 1 hour
  acquisition of peripheral and central photoplethysmographic signals with radial, brachial, carotid and femoral sensors
inductive plethysmography | 1 hour
  acquisition of abdominal and thoracic section variations with an inductive plethysmographic vest

SECONDARY OUTCOMES:
link between peripheral and central pulse wave velocity | 1 hour
  Assesment of the link between peripheral and central vascular function with statistical analysis (Linear regression, Bland and Altman test)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane TANGUY, Principal Investigator — University Grenoble Alpes
Locations (1):
- Laboratoire TIMC, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diaz A, Galli C, Tringler M, Ramirez A, Cabrera Fischer EI. Reference values of pulse wave velocity in healthy people from an urban and rural argentinean population. Int J Hypertens. 2014;2014:653239. doi: 10.1155/2014/653239. Epub 2014 Aug 24. PMID 25215227
- [Background] Fontecave-Jallon J, Tanguy S. Inductive Plethysmography for aortic Pulse Wave Velocity. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:2711-2714. doi: 10.1109/EMBC44109.2020.9175329. PMID 33018566
- [Background] Fortier C, Agharazii M. Arterial Stiffness Gradient. Pulse (Basel). 2016 Apr;3(3-4):159-66. doi: 10.1159/000438852. Epub 2015 Sep 2. PMID 27195235
- [Background] Fortier C, Sidibe A, Desjardins MP, Marquis K, De Serres SA, Mac-Way F, Agharazii M. Aortic-Brachial Pulse Wave Velocity Ratio: A Blood Pressure-Independent Index of Vascular Aging. Hypertension. 2017 Jan;69(1):96-101. doi: 10.1161/HYPERTENSIONAHA.116.08409. Epub 2016 Nov 7. PMID 27821616
- [Background] Heffernan KS, Stoner L, London AS, Augustine JA, Lefferts WK. Estimated pulse wave velocity as a measure of vascular aging. PLoS One. 2023 Jan 26;18(1):e0280896. doi: 10.1371/journal.pone.0280896. eCollection 2023. PMID 36701358
- [Background] Yu S, McEniery CM. Central Versus Peripheral Artery Stiffening and Cardiovascular Risk. Arterioscler Thromb Vasc Biol. 2020 May;40(5):1028-1033. doi: 10.1161/ATVBAHA.120.313128. Epub 2020 Mar 19. PMID 32188277
- [Background] Weber T, Wassertheurer S, Hametner B, Parragh S, Eber B. Noninvasive methods to assess pulse wave velocity: comparison with the invasive gold standard and relationship with organ damage. J Hypertens. 2015 May;33(5):1023-31. doi: 10.1097/HJH.0000000000000518. PMID 25668350
- [Background] Wang J, Jing C, Hu X, Cui J, Tang Q, Tu L, Zhao S, Huang J, Guo D, Li Y, Xu J. Assessment of aortic to peripheral vascular stiffness and gradient by segmented upper limb PWV in healthy and hypertensive individuals. Sci Rep. 2023 Nov 13;13(1):19859. doi: 10.1038/s41598-023-46932-0. PMID 37963909
- [Background] Townsend RR, Wilkinson IB, Schiffrin EL, Avolio AP, Chirinos JA, Cockcroft JR, Heffernan KS, Lakatta EG, McEniery CM, Mitchell GF, Najjar SS, Nichols WW, Urbina EM, Weber T; American Heart Association Council on Hypertension. Recommendations for Improving and Standardizing Vascular Research on Arterial Stiffness: A Scientific Statement From the American Heart Association. Hypertension. 2015 Sep;66(3):698-722. doi: 10.1161/HYP.0000000000000033. Epub 2015 Jul 9. No abstract available. PMID 26160955
- [Background] Sztrymf B, Jacobs F, Chemla D, Richard C, Millasseau SC. Validation of the new Complior sensor to record pressure signals non-invasively. J Clin Monit Comput. 2013 Dec;27(6):613-9. doi: 10.1007/s10877-013-9477-y. Epub 2013 May 17. PMID 23681924
- [Background] Salvi P, Valbusa F, Kearney-Schwartz A, Labat C, Grillo A, Parati G, Benetos A. Non-Invasive Assessment of Arterial Stiffness: Pulse Wave Velocity, Pulse Wave Analysis and Carotid Cross-Sectional Distensibility: Comparison between Methods. J Clin Med. 2022 Apr 15;11(8):2225. doi: 10.3390/jcm11082225. PMID 35456316
- [Background] Salvi P, Lio G, Labat C, Ricci E, Pannier B, Benetos A. Validation of a new non-invasive portable tonometer for determining arterial pressure wave and pulse wave velocity: the PulsePen device. J Hypertens. 2004 Dec;22(12):2285-93. doi: 10.1097/00004872-200412000-00010. PMID 15614022
- [Background] Obeid H, Khettab H, Marais L, Hallab M, Laurent S, Boutouyrie P. Evaluation of arterial stiffness by finger-toe pulse wave velocity: optimization of signal processing and clinical validation. J Hypertens. 2017 Aug;35(8):1618-1625. doi: 10.1097/HJH.0000000000001371. PMID 28379892
- [Background] Karimpour P, May JM, Kyriacou PA. Photoplethysmography for the Assessment of Arterial Stiffness. Sensors (Basel). 2023 Dec 17;23(24):9882. doi: 10.3390/s23249882. PMID 38139728